CLINICAL TRIAL: NCT04800328
Title: Reliability of Infant Neurological International Battery (INFANIB) Among Hospitalized Preterm Infants.
Brief Title: How Accurate INFANIB is Among Hospitalized Preterm Infants
Status: Completed | Type: Observational
Sponsor: Asir John Samuel (Other)
Collaborators: Maharishi Markendeswar University (Deemed to be University) (Other)
Responsible Party: Sponsor-Investigator, Asir John Samuel, Associate Professor, Maharishi Markandeshwar Institute of Physiotherapy and Rehabilitation, Maharishi Markendeswar University (Deemed to be University)
Organization: Maharishi Markendeswar University (Deemed to be University) (Other)
Other Study IDs: MMDU/IEC/1835
Record Dates: First submitted 2021-03-09; First posted 2021-03-16 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Preterm Infants
Keywords: Neonatal; Preterm; NICU; Newborn; INFANIB
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Reliability of infant neurological international battery (INFANIB) among hospitalized preterm infants will be checked. This study will mainly focus on test-retest reliability.

DETAILED DESCRIPTION:
Background: NICU is a specialised intensive care unit that treats and cares for premature or critically ill newborn babies. A special category of high-risk babies consists of premature infants. Their motor growth differs from that of healthy full-term infants and their occurrence of motor disorders is greater. The outcome of neuromotor disorders can be substantially changed by treatments during the first year of life. So in order to detect these neuromotor disorder there must be a reliable screening tool present. Hence, in this study we will check reliability of INFANIB.

Purpose: Reliability of INFANIB among hospitalized preterm infants. Methodology: It will be an observational study and will be carried out in Neonatal Intensive Care Unit (NICU). The study will recruit preterm infants that are stable and are present without any respiratory assistive devices.

INFANIB screening tool will be performed on these infants. It has 20 items that measure the state of the infant for body tone and posture, primitive reflexes and French angles in the supine, prone, sitting, standing and suspended position upto 18 months. But we will take only preterm infants so only 14 items will be assessed and infants will be scored accordingly. The main focus will be on test- retest reliability.

Discussion: A similar research has been carried out in Iran and China, that established that reliability of INFANIB is excellent. Another research was carried out in India that stated INFANIB's reliability to be low. So this study is required to be carried out in India to know the actual results.

ELIGIBILITY:
Inclusion Criteria:

1. Preterm neonates.
2. Stable neonates.

Exclusion Criteria:

1. Unstable neonates.
2. Neonates on respiratory assistive devices.

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Stable preterm infants admitted in Neonatal intensive care unit.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-04-10 (Actual)

PRIMARY OUTCOMES:
INFANIB score | Change from score of INFANIB scale at three consecutive days.
  Measuring neurodevelopmental maturity among neonates

CONTACTS AND LOCATIONS:
Overall Officials: Asir J Samuel, MPT, PhD, Study Chair — Maharishi Markandeshwar Institute of Physiotherapy and Rehabilitation; Dimple Thapar, BPT, Principal Investigator — Maharishi Markandeshwar Institute of Physiotherapy and Rehabilitation
Locations (1):
- Neonatal Intensive Care Unit, Maharishi Markandeshwar Hospital, Ambāla, Haryana, India